CLINICAL TRIAL: NCT06984393
Title: Tele-Rehabilitation Intervention in Community-Based Healthcare for Patients With Parkinson's Disease (DHEAL-COM-PD)
Acronym: DHEAL-COM-PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: INRCA_007_2024
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease; Older People
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Older peple with Parkinson disease
  Interventions: Other: home tele-rehabilitation
- Usual care (Sham Comparator): Older peple with Parkinson disease
  Interventions: Other: Usual care

INTERVENTIONS:
Other: home tele-rehabilitation — Patients will receive a personalised home tele-rehabilitation exercise program consisting of 3 sessions per week for a duration of 12 weeks. The sessions will be organised as follows: one session will be conducted via tele-rehabilitation with the support of a physiotherapist in small groups of up to 5 patients; in the remaining two sessions, the patient will perform the exercises independently at home. BTS TELEREHAB is the platform that will allow the delivery of remote rehabilitation services. The patient is given the system to take home, where they will connect the small Brain PC, that is the computer unit of the BTS TELEREHAB solution, to their television. Before starting the rehabilitation program, the patient will receive training with the technology in the hospital, in the presence of the physiotherapist. During motor rehabilitation sessions, the patient wears a special inertial sensor, the G-Sensor device.
  Arms: Intervention arm
Other: Usual care — Participants will receive a booklet containing information and activities on well-being. They will be invited to do whatever they wish with the information booklet and the proposed exercises.
  Arms: Usual care

SUMMARY:
The study aims to measure the improvement in functional capacity in a group of elderly people suffering from early-stage Parkinson's disease (Hoehn & Yahr scale 1-3), following a telerehabilitation intervention integrated with BTS TELEREHAB technology.

DETAILED DESCRIPTION:
The DHEAL-COM-PD project aims to evaluate the improvement in physical performance of Parkinson's disease patients following an integrated rehabilitation intervention with technology in telerehabilitation. In fact, the project involves the administration of a rehabilitation intervention in telerehabilitation integrated with BTS TELEREHAB technology, which is able to recognize the patient's movements and analyze them according to quantitative (repetitions) and qualitative (postural and balance)-indicators.

The trial is a feasibility study, with single-blind randomized controlled trial type experimental design. Forty older adults with Parkinson's disease will be recruited for the study and randomized into two groups: the experimental group, that will perform tele-rehabilitation at home with a non-immersive virtual reality system, and the control group. Patients in the control group will be offered activities to perform at home, with the same frequency, in line with the usual care activities already proposed by the Rehabilitation Unit.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from Parkinson's disease: Hoehn & Yahr stage I-III;
* Functional Ambulation Category (FAC) score ≥ 3;
* Stability of drug treatment for at least 1 month;
* Maintaining an upright position independently > 30";
* No acute or untreated health problems;
* Mini Mental State Examination (MMSE) ≥ 24;
* Geriatric Depression Score (GDS) < 2;

Exclusion Criteria:

* Myocardial infarction or stroke within 6 months;
* Painful arthritis, spinal stenosis, amputation, painful foot lesions, or neuropathy that limits balance and mobility;
* Uncontrolled hypertension
* Metastatic cancer or immunosuppressive therapy;
* Significant visual or hearing impairment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-02 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in physical performance | at baseline and 12 weeks later
  Physical performance will be evaluated by the Performance-Oriented Mobility Assessment (POMA) test. The total POMA (POMA-T) consists of two sub-scales: the balance rating scale ("balance scale" or POMA-B) and the gait rating scale ("gait scale" or POMA-G). The POMA-B assesses the subject through postures and changes in position that reflect stability patterns related to activities of daily living. In the POMA-G, qualitative aspects of locomotion are considered instead. Each item is scored based on a two- or three-point scale, with a maximum score (POMA-T), derived from the sum of the two sub-scales, of 28 points: in detail, the maximum score for POMA-B is 16, while for POMA-G the maximum score is 12.

SECONDARY OUTCOMES:
Symptoms of Parkinson's disease progression | at baseline and 12 weeks later
  The Symptoms of Parkinson's disease will be evaluated by the Hoen & Yahr Scale. The stages of the scale are: 1 - Unilateral involvement only; 1.5 - Unilateral and axial involvement; 2 - Bilateral involvement without impairment of balance; 2.5 - Mild bilateral involvement without recovery on the pull test; 3 - Mild to moderate bilateral involvement; postural instability; physically self-sufficient; 4 - Severe disability; still able to walk or stand without assistance; 5 - Bedridden or wheelchair-bound.
Improvement in lower limb function | at baseline and 12 weeks later
  It will be measured by the Short Physical Performance Battery (SPPB). The total scale score has a range from 0 to 12, with 12 indicating the maximum performance.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Bevilacqua, PhD, Study Director — IRCCS INRCA, Ancona, Italy
Locations (1):
- IRCCS INRCA Hospital, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No